CLINICAL TRIAL: NCT03996044
Title: Comparative Study Between Photodynamic Therapy Using Urucum + LED and Probiotics in Halitosis Reduction - Controlled Clinical Trial
Brief Title: Comparative Study Between Photodynamic Therapy With Urucum and LED and Probiotics in Halitosis Reduction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pamella
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Halitosis
MeSH Terms: conditions — Halitosis | interventions — Probiotics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Thirteen patients who will receive treatment with teeth brushing, dental floss and tongue scraper.
  Interventions: Other: Teeth brushing and flossing; Other: Tongue scraping
- Group 2 (Experimental): Thirteen patients who will receive treatment with teeth brushing, dental floss and antimicrobial photodynamic therapy applied to the back and middle third of the tongue.
  Interventions: Other: Teeth brushing and flossing; Radiation: Antimicrobial Photodynamic Therapy (aPDT)
- Group 3 (Experimental): Thirteen patients who will receive treatment with teeth brushing, dental floss and probiotics.
  Interventions: Other: Teeth brushing and flossing; Biological: Probiotics
- Group 4 (Experimental): Thirteen patients who will receive treatment with teeth brushing, dental floss, antimicrobial photodynamic therapy applied to the back and middle third of the tongue and probiotics..
  Interventions: Other: Teeth brushing and flossing; Radiation: Antimicrobial Photodynamic Therapy (aPDT); Biological: Probiotics

INTERVENTIONS:
Other: Teeth brushing and flossing — All participants will be instructed to brush with dentifrice containing amine fluoride in their composition (Elmex®) and floss with dental flossing, 3 times a day after meals for 30 days.
Other: Tongue scraping — Tongue scraping will be performed by the same operator on all participants. Posterior-anterior movements will be performed with the scraper over the tongue dorsum, followed by cleaning the scraper with a gauze. This procedure will be performed ten times in each patient, in order to standardize the mechanical removal of the tongue coating.
  Arms: Group 1
Radiation: Antimicrobial Photodynamic Therapy (aPDT) — One session of aPDT will be performed with the photosensitizer (PS) urucum manipulated at a concentration of 20% (Fórmula e Ação®) in spray, to be applied in sufficient quantity to cover the middle third and back of the tongue (5 sprinkles) for 5 minutes for incubation. The excess will be removed with a sucker in order to keep the surface wet with the PS itself, without using water. Six points with a distance of 1 cm between them will be irradiated, considering the halo of light scattering and effectiveness of aPDT. The apparatus shall be precalibrated at wavelength 440-480nm for 60 seconds per point, irradiance of 450mW/cm and the light shall be irradiated so that a halo of 2cm diameter is formed per point.
  Arms: Group 2; Group 4
Biological: Probiotics — Pharmacy-manipulated capsules containing strains of Lactobacillus salivarius WB21 (6.7 x 108 CFU) and xylitol (280mg) will be used. Forty-two capsules will be delivered for each patient, who should take 1 capsule 3 times a day after meals for 14 days.
  Arms: Group 3; Group 4

SUMMARY:
Introduction: Halitosis is a term that defines any foul odor emanating from the oral cavity. The origin may be local or systemic. The aim of the proposed project is to determine whether treatment with antimicrobial photodynamic therapy (aPDT) and treatment with probiotics are effective at eliminating halitosis. Methods and analysis: Fifty-two patients from 18 to 25 years old with a diagnosis of halitosis (H2S≥112 ppb determined by gas chromatography) will be randomly allocated to four groups (n=13) who will receive different treatments: Group 1 - treatment with teeth brushing, dental floss and tongue scraper; Group 2 - brushing, dental floss and aPDT; Group 3 - brushing, dental floss and probiotics; Group 4 - brushing, flossing, aPDT and probiotics. The results of the halimeter testing will be compared before, immediately after, seven days and thirty days after treatment. The microbiological analysis of the coated tongue will be performed at these same times. The quantitative analysis will be conducted using real-time PCRq. The normality of the data will be determined using the Shapiro-Wilk test. Data with normal distribution will be analyzed using analysis of variance (ANOVA). Non-parametric data will be analyzed using the Kruskal-Wallis test. The Wilcoxon test will be used to analyze the results of each treatment at the different evaluation periods. Ethics and dissemination: This study has been approved by the Ethics Committee of UNINOVE under process number 3.669.442. Results will be published in peer-reviewed journals and will be presented at national and international conferences.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 25 years;
* Sulphide (SH2) ≥ 112 ppb in the gas chromatography.

Exclusion Criteria:

* Dentofacial anomalies (such as cleft lip and cleft palate);
* Undergoing orthodontic and/or orthopedic treatment;
* Undergoing oncological treatment;
* Systemic alterations (gastrointestinal, renal, hepatic);
* Treatment with antibiotics up to 1 month before the survey;
* Pregnant.
* Individuals with fissured tongue

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change in halimetry (gas chromatography) | Baseline, immediately after treatment, 7 days and 30 days after treatment.
  Oral air collection will follow the manufacturer's guidelines (Oral ChromaTM Manual Instruction) where the participant will be instructed to rinse with cysteine (10 mM) for 1 minute, then remain with his/her mouth closed for 1 minute. A syringe from the same manufacturer for collection of mouth air will be introduced into the patient's mouth. During 1 minute the patient will remain closed mouth, breathing through the nose, without touching the syringe with the tongue. The plunger will be pulled out, we will re-empty the syringe air into the patient's mouth and again pull the plunger to fill the syringe with the breath sample. We will wipe the tip of the syringe with gauze to remove moisture from the saliva, place the gas injection needle in the syringe, and adjust the plunger to 0.5 ml. The gases collected at the entrance door of the appliance are injected in a single movement.

SECONDARY OUTCOMES:
Change in microbiological analysis of tongue coating | Baseline, immediately after treatment, 7 days and 30 days after treatment.
  Samples of the tongue coating will be collected using a sterile swab that will be passed on the surface of the back of the tongue with a back and forth movement (10 times). Samples will be deposited in sterile tubes that will be identified and stored at -80°C until analyzed. After thawing, the samples will be vortexed for one minute. For extraction of bacterial DNA, samples will be boiled for 10 minutes and then centrifuged at 10,000 rpm for 10 minutes. The supernatant will be placed in a new microtube containing 100μL of phenol/chloroform/isoamyl alcohol (25: 24: 1), followed by ethanol precipitation. The purified DNA will be resuspended in TE buffer. The levels of P. gingivalis, T. forsythia and T. denticola, will be analyzed by quantitative PCR. The quantitative analysis will be performed using real-time PCR using Step One Plus Thermal-Time PCR System and fluorescence-detected products using the Quantimix Easy SYG Kit, following the protocol recommended by the manufacturer.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Nove de Julho, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Motta PB, Goncalves MLL, Gallo JMAS, Sobral APT, Motta LJ, Mayer MPA, Kawamoto D, de Andrade DC, Santos EM, Fernandes KPS, Mesquita-Ferrari RA, Deana AM, Horliana ACRT, Kalil Bussadori S. Short term effect of antimicrobial photodynamic therapy and probiotic L. salivarius WB21 on halitosis: A controlled and randomized clinical trial. PLoS One. 2024 Jul 2;19(7):e0297351. doi: 10.1371/journal.pone.0297351. eCollection 2024. PMID 38954692
- [Derived] Motta PB, Motta LJ, Costa da Mota AC, Leal Goncalves ML, Silva T, Momolli M, de Andrade DC, Santos Fernandes KP, Mesquita-Ferrari RA, Deana AM, Wainwright M, Prates RA, Horliana ACRT, Bussadori SK. Comparative study between photodynamic therapy with urucum + Led and probiotics in halitosis reduction-protocol for a controlled clinical trial. PLoS One. 2021 May 14;16(5):e0247096. doi: 10.1371/journal.pone.0247096. eCollection 2021. PMID 33989296